CLINICAL TRIAL: NCT03474367
Title: Cost-effectiveness of Urgent-start Therapies Hemodialysis and Peritoneal Dialysis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Alexandre Minetto Brabo, Mastering Student, Universidade Estadual Paulista Júlio de Mesquita Filho
Other Study IDs: 97/2017
Record Dates: First submitted 2017-06-28; First posted 2018-03-22 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Cost-effectiveness Analysis; Chronic Kidney Disease Requiring Chronic Dialysis
Keywords: Unplanned Peritoneal Dialysis; Unplanned Hemodialysis; Cost-Benefit Analysis; Dialysis; Peritoneal Dialysis; Hemodialysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Unplanned Peritoneal Dialysis: CKD patients stage 5 (eGFR < 15 ml/min/1,73m²) or stages 4 with abrupt worsening renal function requiring dialysis treatment immediately, followed or not by nephrologists prior to renal replacement therapy (RRT) indication, that agree to initiate peritoneal dialysis (PD) in less than 48 hours after implantation of the peritoneal catheter, without family training or adequacy of the home. The patient must not have any absolute contraindications to initiate PD, which include: presence of recent abdominal surgery (less than 30 days); multiple previous abdominal surgery (more than two); presence of fibrosis or peritoneal adhesions; fungal peritonitis; severe respiratory insufficiency (FiO2> 70%); abdominal infections; severe hyperkalemia with changes characteristic in ECG; and acute pulmonary edema. These patients will be treated with HD.
- Unplanned Hemodialysis: CKD patients stage 5 (eGFR < 15 ml/min/1,73m²) or stages 4 with abrupt worsening renal function requiring dialysis treatment immediately, followed or not by nephrologists prior to renal replacement therapy (RRT) indication, that agree to initiate HD without a functional arteriovenous fistula, ie, with a central venous catheter (nontunneled or tunneled).

SUMMARY:
This study will evaluate the cost-effectiveness of unplanned dialysis (peritoneal dialysis and hemodialysis) in chronic kidney disease (CKD) during the first year of therapy in a single center.

DETAILED DESCRIPTION:
Despite evidence of worse outcomes, initiation of renal replacement therapy by unplanned modalities in chronic kidney disease (CKD) patients is the reality in the practice for both hemodialysis and peritoneal dialysis. Unplanned therapy peritoneal dialysis (PD) is the initiation of the modality in less than 48 hours after implantation of the peritoneal catheter, without family training or adequacy of the home. Unplanned hemodialysis (HD) is the initiation of the method without a functional arteriovenous fistula, i.e., with a central venous catheter (nontunneled or tunneled).

Growing evidence shows unplanned PD (or urgent start PD) as a viable and safe alternative to unplanned HD, with the similar rates of infection and survival.

On planned scenario, solid studies demonstrate that PD has a better cost-effectiveness when compared to HD, however the literature lacks in this kind of analysis in unplanned methods.

Briefly, the workgroup will follow patients that would anyway start a Renal Replacement Therapy by an unplanned method and register Government payment for the therapy, including the therapy direct costs and the costs with events (internation, infection), access for dialysis, laboratory and CKD specific medications to performed a cost-effectiveness analysis in both groups (Unplanned Hemodialysis and Unplanned Peritoneal Dialysis).

The workgroup is responsible for the placement of the catheters (PD and HD) using the Seldinger Technique.

The study is unicentric, the therapy is continuous and necessary for the maintenance of life; therefore, no great difficult in the follow up is expected. A database with up-to-date information of patients will be functional during the study.

A Markov model will be developed to assess the relative cost-effectiveness of different dialysis modality distribution scenarios versus current practice. The model considers a hypothetical adult incident patient cohort with end-stage renal disease (ESRD) requiring dialysis and adopts payer perspective. Markov models have been used to model dialysis treatment in previous economic analyses and are widely accepted to be suitable for modelling chronic condition

Statistical analysis plan:

From the study protocol, the data will be entered in a spreadsheet and verified typographical errors and their analysis will be performed using the statistical program Statistical Analysis System (SAS) for Windows (version 9.2: SAS Institute, Cary, North Carolina, USA, 2012).

Considering an alpha error of 0.05 and a beta error of 0.2, power of statistic test of 0.8 and cost difference detection between groups of 15%, the calculated sample size for each group is 94 patients.

Initially descriptive analysis will be done for all patients treated in the period, calculated measures of central tendency and dispersion for continuous variables and frequencies for categorical variables.

For the analysis of repeated measures, asymmetric distribution (gamma) under the Generalized Linear Model (GENMOD) procedure will be used.

Chi Square will be used to compare categorical variable between the two groups. T test or Mann-Whitney will be used to compare parametric continue variables.

By the utilization of Kaplan Meyer and log rank, survival curves of the two groups will be presented at the end of the study. A p-value of 5% or lower will be considered to be statistically significant

ELIGIBILITY:
Inclusion Criteria:

* Ambulatorial Chronic Kidney Disease patients stage 5 (eGFR < 15 ml/min) or stages 4 with abrupt worsening requiring dialysis treatment immediately followed or not by nephrologists prior to Renal Replacement Therapy indication.

Exclusion Criteria:

* Transitions between HD and PD
* Patients with functional arteriovenous fistula entering hemodialysis
* Patients with functional PD access implanted ate least 48h before the first use
* Patient or family trained in PD and/or with the right adequacy of the home

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Incident dialysis patients.
Sampling Method: Non-Probability Sample
Enrollment: 198 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-03-12 (Estimated); Study Completion 2021-12-12 (Estimated)

PRIMARY OUTCOMES:
Cost effectiveness analysis of unplanned PD and HD at the General Hospital of the School of Medicine of Botucatu (HC-FMB) | 12 months
  Cost effectiveness analysis of unplanned PD and HD with the data collected at our center

SECONDARY OUTCOMES:
Cost effectiveness analysis of unplanned PD and HD in national and international scenario | 12 months
  Transpose the cost-effectiveness analysis to a national and international scenario, using a Markov model

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina de Botucatu, Botucatu, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Woo KT, Choong HL, Wong KS, Tan HB, Chan CM. The contribution of chronic kidney disease to the global burden of major noncommunicable diseases. Kidney Int. 2012 May;81(10):1044-1045. doi: 10.1038/ki.2012.39. No abstract available. PMID 22543907
- [Background] Eggers PW. Has the incidence of end-stage renal disease in the USA and other countries stabilized? Curr Opin Nephrol Hypertens. 2011 May;20(3):241-5. doi: 10.1097/MNH.0b013e3283454319. PMID 21422925
- [Background] Klarenbach SW, Tonelli M, Chui B, Manns BJ. Economic evaluation of dialysis therapies. Nat Rev Nephrol. 2014 Nov;10(11):644-52. doi: 10.1038/nrneph.2014.145. Epub 2014 Aug 26. PMID 25157840
- [Background] Haller M, Gutjahr G, Kramar R, Harnoncourt F, Oberbauer R. Cost-effectiveness analysis of renal replacement therapy in Austria. Nephrol Dial Transplant. 2011 Sep;26(9):2988-95. doi: 10.1093/ndt/gfq780. Epub 2011 Feb 10. PMID 21310740
- [Background] Howard K, Salkeld G, White S, McDonald S, Chadban S, Craig JC, Cass A. The cost-effectiveness of increasing kidney transplantation and home-based dialysis. Nephrology (Carlton). 2009 Feb;14(1):123-32. doi: 10.1111/j.1440-1797.2008.01073.x. PMID 19207859
- [Background] Korevaar JC, Feith GW, Dekker FW, van Manen JG, Boeschoten EW, Bossuyt PM, Krediet RT; NECOSAD Study Group. Effect of starting with hemodialysis compared with peritoneal dialysis in patients new on dialysis treatment: a randomized controlled trial. Kidney Int. 2003 Dec;64(6):2222-8. doi: 10.1046/j.1523-1755.2003.00321.x. PMID 14633146
- [Background] Vonesh EF, Snyder JJ, Foley RN, Collins AJ. Mortality studies comparing peritoneal dialysis and hemodialysis: what do they tell us? Kidney Int Suppl. 2006 Nov;(103):S3-11. doi: 10.1038/sj.ki.5001910. PMID 17080109
- [Background] Perl J, Wald R, McFarlane P, Bargman JM, Vonesh E, Na Y, Jassal SV, Moist L. Hemodialysis vascular access modifies the association between dialysis modality and survival. J Am Soc Nephrol. 2011 Jun;22(6):1113-21. doi: 10.1681/ASN.2010111155. Epub 2011 Apr 21. PMID 21511830
- [Background] Heaf JG, Lokkegaard H, Madsen M. Initial survival advantage of peritoneal dialysis relative to haemodialysis. Nephrol Dial Transplant. 2002 Jan;17(1):112-7. doi: 10.1093/ndt/17.1.112. PMID 11773473
- [Background] Termorshuizen F, Korevaar JC, Dekker FW, Van Manen JG, Boeschoten EW, Krediet RT; Netherlands Cooperative Study on the Adequacy of Dialysis Study Group. Hemodialysis and peritoneal dialysis: comparison of adjusted mortality rates according to the duration of dialysis: analysis of The Netherlands Cooperative Study on the Adequacy of Dialysis 2. J Am Soc Nephrol. 2003 Nov;14(11):2851-60. doi: 10.1097/01.asn.0000091585.45723.9e. PMID 14569095
- [Background] Dias DB, Banin V, Mendes ML, Barretti P, Ponce D. Peritoneal dialysis can be an option for unplanned chronic dialysis: initial results from a developing country. Int Urol Nephrol. 2016 Jun;48(6):901-6. doi: 10.1007/s11255-016-1243-x. Epub 2016 Feb 20. PMID 26897038
- [Background] Silva TN, de Marchi D, Mendes ML, Barretti P, Ponce D. Approach to prophylactic measures for central venous catheter-related infections in hemodialysis: a critical review. Hemodial Int. 2014 Jan;18(1):15-23. doi: 10.1111/hdi.12071. Epub 2013 Aug 14. PMID 23944971
- [Background] Mendes ML, Castro JH, Silva TN, Barretti P, Ponce D. Effective use of alteplase for occluded tunneled venous catheter in hemodialysis patients. Artif Organs. 2014 May;38(5):399-403. doi: 10.1111/aor.12186. Epub 2013 Oct 3. PMID 24117542
- [Background] Koch M, Kohnle M, Trapp R, Haastert B, Rump LC, Aker S. Comparable outcome of acute unplanned peritoneal dialysis and haemodialysis. Nephrol Dial Transplant. 2012 Jan;27(1):375-80. doi: 10.1093/ndt/gfr262. Epub 2011 May 28. PMID 21622993
- [Background] Lobbedez T, Lecouf A, Ficheux M, Henri P, Hurault de Ligny B, Ryckelynck JP. Is rapid initiation of peritoneal dialysis feasible in unplanned dialysis patients? A single-centre experience. Nephrol Dial Transplant. 2008 Oct;23(10):3290-4. doi: 10.1093/ndt/gfn213. Epub 2008 Apr 19. PMID 18424817
- [Background] Alkatheeri AM, Blake PG, Gray D, Jain AK. Success of Urgent-Start Peritoneal Dialysis in a Large Canadian Renal Program. Perit Dial Int. 2016 Mar-Apr;36(2):171-6. doi: 10.3747/pdi.2014.00148. Epub 2015 Sep 15. PMID 26374834
- [Background] Povlsen JV. Unplanned start on assisted peritoneal dialysis. Contrib Nephrol. 2009;163:261-263. doi: 10.1159/000223808. Epub 2009 Jun 3. PMID 19494623
- [Background] Chang YT, Hwang JS, Hung SY, Tsai MS, Wu JL, Sung JM, Wang JD. Cost-effectiveness of hemodialysis and peritoneal dialysis: A national cohort study with 14 years follow-up and matched for comorbidities and propensity score. Sci Rep. 2016 Jul 27;6:30266. doi: 10.1038/srep30266. PMID 27461186
- [Background] Atapour A, Eshaghian A, Taheri D, Dolatkhah S. Hemodialysis versus peritoneal dialysis, which is cost-effective? Saudi J Kidney Dis Transpl. 2015 Sep;26(5):962-5. doi: 10.4103/1319-2442.164578. PMID 26354569
- [Background] Liu FX, Ghaffari A, Dhatt H, Kumar V, Balsera C, Wallace E, Khairullah Q, Lesher B, Gao X, Henderson H, LaFleur P, Delgado EM, Alvarez MM, Hartley J, McClernon M, Walton S, Guest S. Economic evaluation of urgent-start peritoneal dialysis versus urgent-start hemodialysis in the United States. Medicine (Baltimore). 2014 Dec;93(28):e293. doi: 10.1097/MD.0000000000000293. PMID 25526471
- [Background] Passadakis PS, Oreopoulos DG. Peritoneal dialysis in patients with acute renal failure. Adv Perit Dial. 2007;23:7-16. PMID 17886595
- [Background] Mowatt G, Vale L, Perez J, Wyness L, Fraser C, MacLeod A, Daly C, Stearns SC. Systematic review of the effectiveness and cost-effectiveness, and economic evaluation, of home versus hospital or satellite unit haemodialysis for people with end-stage renal failure. Health Technol Assess. 2003;7(2):1-174. doi: 10.3310/hta7020. No abstract available. PMID 12773260
- [Background] Kirby L, Vale L. Dialysis for end-stage renal disease. Determining a cost-effective approach. Int J Technol Assess Health Care. 2001 Spring;17(2):181-9. doi: 10.1017/s0266462300105045. PMID 11446130
- [Derived] Htay H, Johnson DW, Craig JC, Teixeira-Pinto A, Hawley CM, Cho Y. Urgent-start peritoneal dialysis versus haemodialysis for people with chronic kidney disease. Cochrane Database Syst Rev. 2021 Jan 27;1(1):CD012899. doi: 10.1002/14651858.CD012899.pub2. PMID 33501650
- [Derived] Htay H, Johnson DW, Craig JC, Teixeira-Pinto A, Hawley CM, Cho Y. Urgent-start peritoneal dialysis versus conventional-start peritoneal dialysis for people with chronic kidney disease. Cochrane Database Syst Rev. 2020 Dec 15;12(12):CD012913. doi: 10.1002/14651858.CD012913.pub2. PMID 33320346
- See also: National Kidney Foundation. 2016 — http://kidney.org/kidneydisease/global-facts-about-kidney-disease
- See also: Danish Nephrology Registry, Annual Report 2011 — http://www.nephrology.dk
- See also: Census of the Brazillian Society of Nephrology 2014 — http://www.sbn.org.br